CLINICAL TRIAL: NCT00567073
Title: A Sub-registry to Observe the Effect of Alglucosidase Alfa or Avalglucosidase Alfa Treatment on Pregnancy and Infant Growth in Women With Pompe Disease
Brief Title: Pompe Pregnancy Sub-Registry
Status: Recruiting | Type: Observational
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: AGLU03506
Record Dates: First submitted 2007-12-01; First posted 2007-12-04 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Glycogen Storage Disease Type II (GSD-II); Pompe Disease (Late-onset); Glycogenesis 2 Acid Maltase Deficiency
Keywords: Glycogen Storage Disease Type II (GSD-II); GSD-II; Pompe Disease; Pompe Disease (Late-Onset); Acid Maltase Deficiency Disease; Glycogenosis II
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Pregnant women with confirmed diagnosis of Pompe Disease: No experimental intervention is given. Pregnant women with confirmed diagnosis of Pompe disease that are participating in the Pompe Registry (NCT00231400) and consented to participate in the Pompe Pregnancy Sub-registry, regardless of whether she is receiving disease-specific therapy (such as ERT with alglusidase alfa or avalglucosidase alfa) and irrespective of the commercial product with which she may be treated.
- Pregnant women receiving no treatment for Pompe disease: Pregnant women with Pompe disease enrolled in the Pompe disease registry (NCT00231400) who are not receiving treatment
- Infants born to mothers receiving treatment for Pompe disease: The infants of mothers with Pompe disease enrolled in the Pompe disease registry (NCT00231400) where the mothers are receiving treatment of alglucosidase alfa (Myozyme/Lumizyme) or avalglucosidase alfa (Nexviadyme/Nexviazyme)
- Infants born to mothers receiving no treatment for Pompe disease: The infants of mothers with Pompe disease enrolled in the Pompe Disease Registry (NCT00231400) where the mothers are not receiving Treatment

SUMMARY:
This Sub-registry is a multicenter, international, longitudinal, observational, and voluntary program designed to track pregnancy outcomes for any pregnant woman enrolled in the Pompe Registry, regardless of whether she is receiving disease-specific therapy (such as ERT with alglucosidase alfa or avalglucosidase alfa) and irrespective of the commercial product with which she may be treated. No experimental intervention is given; thus a patient will undergo clinical assessments and receive standard of care treatment as determined by the patient's physician.

The primary objective of this Sub-registry is to track pregnancy outcomes, including complications and infant growth, in all women with Pompe disease during pregnancy, regardless of whether they receive disease-specific therapy, such as ERT with alglucosidase alfa or avalglucosidase alfa.

DETAILED DESCRIPTION:
Study Design Time Perspective: Retrospective and Prospective

ELIGIBILITY:
Inclusion Criteria:

Eligible women must:

* be enrolled in the Pompe registry (NCT00231400)
* be pregnant, or have been pregnant with appropriate medical documentation available.
* provide a signed informed consent and authorization form(s) to participate in the Sub-Registry prior to any Sub-Registry-related data collection being performed.

Note: It is recommended that pregnancy data be collected on eligible women regardless of infant enrollment. In the event of patients having multiple pregnancies, participation in this Sub-Registry is encouraged for each individual pregnancy.

Exclusion Criteria:

There are no exclusion criteria for this Sub-Registry

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant Females with Pompe disease and/or infants born to females with Pompe disease. Participants may or may not be receiving therapy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2007-06-18 (Actual); Primary Completion 2034-01-31 (Estimated); Study Completion 2034-01-31 (Estimated)

PRIMARY OUTCOMES:
Pregnancy outcomes, including complications and infant growth, in all women with Pompe disease during pregnancy, regardless of whether they receive disease-specific therapy such as ERT with alglucosidase alfa or avalglucosidase alfa | 10 Months
Follow-up of infants born to women with Pompe disease for 3 years post-partum | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Genzyme, a Sanofi Company
Locations (26):
- United States (10):
  - Barrow Neurol Group- Site Number : 840087, Phoenix, Arizona
  - Emory University School Of Medicine- Site Number : 840060, Atlanta, Georgia
  - Indianapolis University School of Medicine- Site Number : 840027, Indianapolis, Indiana
  - Spectrum for Health- Site Number : 840019, Grand Rapids, Michigan
  - New York University School Of Medicine- Site Number : 840040, New York, New York
  - Mt. Sinai School of Medicine- Site Number : 840005, New York, New York
  - Duke University Medical Center Genetics Dept- Site Number : 840037, Durham, North Carolina
  - LSD Data Registry Site LLC- Site Number : 840094, Dublin, Ohio
  - Oregon Health and Science University- Site Number : 840095, Portland, Oregon
  - O&O Alpan, LLC- Site Number : 840025, Fairfax, Virginia
- Investigational Site Number : 056001, Ghent, Belgium
- Croatia (2):
  - Investigational Site Number : 1910001, Zagreb
  - Investigational Site Number : 1910002, Zagreb
- Investigational Site Number : 2030001, Prague, Czechia
- Italy (12):
  - Investigational Site Number : 380008, Brescia
  - Investigational Site Number : 380006, Cagliari
  - Investigational Site Number : 380005, Florence
  - Investigational Site Number : 380004, Genova
  - Investigational Site Number : 380013, Messina
  - Investigational Site Number : 380007, Milan
  - Investigational Site Number : 380009, Monza
  - Investigational Site Number : 380002, Padua
  - Investigational Site Number : 380011, Padua
  - Investigational Site Number : 380003, Pavia
  - Investigational Site Number : 380015, Roma
  - Investigational Site Number : 380012, Roma